CLINICAL TRIAL: NCT06394388
Title: A Cultural Adaptation of the Caregiver TLC Psychoeducational Program to Support Latino Caregivers (CUIDANDO JUNTOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of North Carolina, Charlotte (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julian Montoro, Professor, University of North Carolina, Charlotte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-0291-01; 5P30AG064103 (NIH)
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Caregivers of People With Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental)
  Interventions: Behavioral: Cuidando juntos

INTERVENTIONS:
Behavioral: Cuidando juntos — Caregiver TLC program will be culturally tailored by including a focus on addressing cultural values to promote social connectedness and translated into Spanish (Cuidando Juntos).
  Cuidando Juntos consists of 8 modules: stress management; behavioral activation; building resilience; building self-care skills; managing difficult emotions; reducing isolation; and two on understanding and responding to difficult behaviors of the PLWD.

SUMMARY:
This study will test the feasibility and influence of a behavioral intervention called "Cuidando Juntos" in Latino caregivers of people with dementia. The study will examine if the intervention is well received by Latino caregivers and if the caregivers' social connectedness and loneliness is associated with their levels of stress, burden, and depression.

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaking
* Latino caregivers are those who identify as the primary caregivers of a person with dementia, with whom they co-reside or live close by.
* must have an email address and access to the internet
* Caregivers should report at least a moderate level of stress

Exclusion Criteria:

* None

Min Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Mean change in PHQ-9 to assess depressive symptoms | Baseline to six weeks
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).The scale ranges from 0-27, with higher scores indicating higher depression.
Mean change in Perceived Stress Scale | Baseline to six weeks
  The perceived stress scale is a 4-item questionnaire, with a score range of 0 to 16. Higher scores are correlated with more stress.
Mean change in Zarit Caregiver Burden 6-item version | Baseline to six weeks
  The Zarit caregiver burden 6-item version is a self-administered instrument that ranges from 0-88. Higher scores indicate more burden.
Mean change in Caregiver Self-Efficacy Scale (CSES-8) | Baseline to six weeks
  The caregiver self-efficacy scale is an 8-item scale developed to reflect components of typical caregiver support interventions that range from 0 to 8. Higher scores indicate being more confident.
Mean change in UCLA Loneliness Scale | Baseline to six weeks
  The UCLA loneliness scale is a 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. The scale measures from 0 to 60; higher scores indicate more loneliness.
Mean change in Social Network Scale | Baseline to six weeks
  The Social network scale is a self-report measure of social engagement that includes engagement with family and friends.The Short version, a 6-item scale, is used. The scale ranges from 0 to 35; higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina, Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No